CLINICAL TRIAL: NCT04920968
Title: Efficacy and Safety of Obinutuzumab Versus Rituximab in Combination With Chemotherapy for Adult Patients With Newly Diagnosed CD20-positive Acute Lymphoblastic Leukemia
Brief Title: Obinutuzumab Versus Rituximab for Acute Lymphoblastic Leukemia/PALG ALL7 "OVERALL"
Acronym: OVERALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-NIO-0002
Record Dates: First submitted 2021-04-25; First posted 2021-06-10 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: CD20-positive Acute Lymphoblastic Leukemia
MeSH Terms: interventions — obinutuzumab; Rituximab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Obinutuzumab (Experimental): Patients in reference arm (Arm A) will receive rituximab. Patients in experimental arm (Arm B) will receive obinutuzumab instead of rituximab in the same time-points.
  Interventions: Drug: Obinutuzumab
- Rituximab (Active Comparator): Patients in reference arm (Arm A) will receive rituximab. Patients in experimental arm (Arm B) will receive obinutuzumab instead of rituximab in the same time-points.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Obinutuzumab — Chemotherapy will be conducted according to PALG ALL7 protocol, which is considered a standard of care in Poland. Patients in experimental arm will receive obinutuzumab .Obinutuzumab: 1000 mg i.v. (first infusion divided into 100 mg on d. 1 and 900 mg on d. 2).
  Arms: Obinutuzumab
Drug: Rituximab — Chemotherapy will be conducted according to PALG ALL7 protocol, which is considered a standard of care in Poland.The protocol includes the use of rituximab in combination chemotherapy. Rituximab: 375 mg/m2 intravenously (i.v.)
  Other Names: Activ comparator
  Arms: Rituximab

SUMMARY:
A multicenter, prospective, randomized and controlled study to compare the efficacy and safety of obinutuzumab and rituximab in adult ALL patients with CD20 expression.Study population is 124 patients (62 in each study group).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Newly diagnosed Acute lymphoblastic leukemia with CD20 expression on at least 20% of blasts.
3. Signed written informed consent.
4. Adequate contraception in case of women with child-bearing potential

Exclusion Criteria:

1. Lymphoblastic lymphoma with bone marrow blasts<20%.
2. Patients with a history of chronic myeloid leukemia or other myeloproliferative disease.
3. Major surgery within 4 weeks before enrollment.
4. Impaired cardiac function: ejection fraction <40% on echocardiography, QTc interval > 450 ms on baseline electrocardiogram. Myocardial infarction within 6 months prior to starting study; other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension, uncontrolled arrhythmias).
5. Active infection e.g. hepatitis B virus, hepatitis C virus, human immunodeficiency virus
6. Other concurrent severe and/or uncontrolled medical conditions: patients with another primary malignant disease, except those that do not currently require treatment; acute or chronic liver, pancreatic or severe renal disease; another severe and/or life-threatening medical disease.
7. Serum creatinine > 2 times the upper normal limit of the laboratory, total bilirubin> 2.5 upper normal limit unless related to Acute lymphoblastic leukemia, aspartate aminotransferase or alanine aminotransferase > 5 upper normal limit, unless related to Acute lymphoblastic leukemia
8. Intolerance to treatment with monoclonal antibody.
9. Positive pregnancy test (beta human chorionic gonadotropin) for women of childbearing age.
10. Inability to obtain written informed consent.
11. Inability to comply with regular monitoring.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving complete remission with Minimal Residual Disease level <0.1% of bone marrow cells after one course of induction treatment. | assessed between days 33-34 since start of Induction I

SECONDARY OUTCOMES:
The proportion of patients achieving complete remission with Minimal Residual Disease level <0.01% of bone marrow cells after consolidation. | assessed between days 20-28 since start of last course of consolidation
complete remission rate after Induction I | assessed between days 33-34 since start of Induction I
Overall complete remission | in 24month follow up
Probability of overall survival | in 24 month follow up
Probability of relapse-free survival | in 24 month follow up
Probability of event-free survival | in 24 month follow up
Cumulative incidence of relapse | in 24 month follow up
Rate of adverse events | in 24 month follow up

CONTACTS AND LOCATIONS:
Locations (19):
- Poland (19):
  - Klinika Hematologii z Pododziałem Chorób Naczyń Uniwersyteckiego, Bialystok
  - Oddział Hematologii Onkologicznej Podkarpacki Ośrodek Onkologiczny, Brzozów
  - Klinika Transplantacji Szpiku i Onkohematologii Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie Państwowy Instytut Badawczy, Oddział w Gliwicach, Gliwice
  - Klinika Hematologii i Transplantacji Szpiku, Samodzielny Publiczny Szpital Kliniczny, Katowice
  - Klinika Hematologii i Transplantacji Szpiku, Świętokrzyskie Centrum Onkologii, Kielce
  - Oddział Hematologii i Chorób Wewnętrznych z Pododdziałem Dziennym Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie Sp. z o.o., Krakow
  - Oddział Hematologiczny Wojewódzkiego Szpitala Specjalistycznego w Legnicy, Legnica
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz
  - Klinika Hematoonkologii I Transplantacji Szpiku, Uniwersytet Medyczny w Lublinie, Lublin
  - Oddział Hematologii i Transplantacji Szpiku Centrum Onkologii Ziemi Lubelskiej im. Św. Jana z Dukli w Lublinie, Lublin
  - Oddział Kliniczny Hematologii Samodzielnego Publicznego Zakładu Opieki Zdrowotnej MSWiA z Warmińsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Klinika Hematologii i Chorób Rozrostowych Układu Krwiotwórczego Uniwersytetu Medycznego w Poznaniu, Poznan
  - Klinika Hematologii Pomorskiego Uniwersytetu Medycznego, Szczecin
  - Oddział Hematologii, Specjalistyczny Szpital Miejski, Torun
  - Klinika Chorób Wewnętrznych i Hematologii Wojskowy Instytut Medyczny, Warsaw
  - Klinika Hematologii, Instytut Hematologii i Transfuzjologii, Warsaw
  - Klinika Hematologii, Onkologii i Chorób Wewnętrznych Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Katedra i Klinika Hematologii, Nowotworów Krwi i Transplantacji Szpiku, Wroclaw
  - Oddział Hematologiczny Z Oddziałem Nowotworów Krwi Dolnośląskie Centrum Transplantacji Komórkowych Z Krajowym Bankiem Dawców Szpiku, Wroclaw